CLINICAL TRIAL: NCT04981886
Title: Intraocular Pressure Reduction Efficacy of Rhopressa and Lumigan in Normal Tension Glaucoma
Acronym: NTG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMS1311
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Normal Tension Glaucoma
Keywords: Glaucoma; Normal tension glaucoma; Intraocular pressure; Central corneal thickness; Corneal hysteresis; Prostaglandin analog; Prostamide
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Normal tension glaucoma subjects with thin corneas (Experimental): NTG subjects with CCT ≤ 540 nm will be randomized to receive either netarsudil or bimatoprost.
  Interventions: Drug: Netarsudil Ophthalmic; Drug: Bimatoprost Ophthalmic
- Group 2: Normal tension glaucoma subjects with thick corneas (Experimental): NTG subjects with CCT > 540 nm will be randomized to receive either netarsudil or bimatoprost.
  Interventions: Drug: Netarsudil Ophthalmic; Drug: Bimatoprost Ophthalmic

INTERVENTIONS:
Drug: Netarsudil Ophthalmic — Subjects will be randomly assigned to this group
  Other Names: Rhopressa
Drug: Bimatoprost Ophthalmic — Subjects will be randomly assigned to this group
  Other Names: Lumigan

SUMMARY:
Glaucoma is the second leading cause of blindness and the first leading cause of irreversible vision loss worldwide. The intraocular pressure (IOP) is the only modifiable risk factor for all the spectrum of glaucoma. Reducing IOP in glaucoma increases the likelihood of preventing progression of the disease and preserving the quality of life of the patient. Although prostaglandin analogs (PGAs) and prostamides (PMs) are de facto first-line treatment options for managing glaucoma, it is a common clinical experience to see their treatment effects plateau to a level beyond which no clinically significant IOP reduction is likely. It is also common to find minimal IOP treatment effects in the following conditions: patients with normal tension glaucoma (NTG), patients with thicker central corneal thickness (CCT), and patients with higher levels of corneal hysteresis (CH). CH is a possible proxy for the ability of the scleral tissue around the optic nerve to dissipate energy away from the optic nerve fibers. Netarsudil, a rho-kinase inhibitor was recently approved by the FDA for the treatment of glaucoma and ocular hypertension. There is a paucity of research on the efficacy of netarsudil in patients with NTG, thicker CCT, and higher levels of CH. This study aims to investigate the above issues by evaluating the efficacy of netarsudil and bimatoprost in subjects with NTG, thicker corneas, and higher levels of CH.

Hypotheses

* Netarsudil will have non-inferior efficacy compared to Bimatoprost in treating NTG.
* Corneal thickness and corneal hysteresis will reduce the efficacy of netarsudil similar to bimatoprost in NTG.
* Netarsudil will change corneal thickness and corneal hysteresis similar to bimatoprost in NTG.

DETAILED DESCRIPTION:
CHARACTERISTICS OF THE SUBJECT POPULATION

1. Target Accrual. The target number of participants we aim to recruit is one hundred and fifteen (115). Participants will be recruited from the patient base of Roberts Eyecare Associates in Vestal, New York, and from referrals from other practices.
2. Gender of the Subjects. There will be no gender restriction in the study.
3. Age Range of Adult Subjects. The age range of participants is 21 to 89 years. This age range is based on the Collaborative Normal Tension Glaucoma Study (CNTGS).
4. Age Range of Pediatric Subjects. Not applicable.
5. Racial and Ethnic Origin. There will be no restriction based on race or ethnicity.
6. Vulnerable Subjects. It is not anticipated that the study will include vulnerable subjects like pregnant persons, breastfeeding persons, persons considering becoming pregnant, children, prisoners, individuals with impaired decision-making capacity, Salus employees and/or students. However, if any subject meeting the inclusion criteria is determined to be a vulnerable subject as defined above, they will be excluded for participation.

METHODS AND PROCEDURES

1. Patient History

   The initial examination will include a comprehensive patient history that will include the following:
   * date of birth
   * race/ethnicity
   * ocular and general medical history
   * list of the medications
   * family ocular and general medical history
   * allergy history
   * social history, including history of smoking, alcohol, and recreational drug use.
2. Procedures at first visit

   1. Ocular Response Analyzer (ORA: Reichert ophthalmic instrument, Buffalo, NY, USA):

      This test will be used to automatically measure corneal hysteresis (CH), corneal corrected intraocular pressure (IOPcc), and Goldman equivalent intraocular pressure (IOPg). At least 5 readings will be taken and the highest 3 wave score readings above 6.5 will be averaged to get measurements for CH, CRF, IOPcc, and IOPg.
   2. Humphrey's Threshold Visual field test:

      The 24-2 threshold Humphrey's visual field analyzer with the sita standard algorithm will be used to determine the status of visual field for all participants. Three visual field tests will be conducted to ensure reliability and repeatability. Visual field test results with > 33% fixation losses, > 33% false positive, or 33% false negative errors will be excluded.
   3. Spectral-Domain Optical Coherence Tomography (SD-OCT) Test The SD-OCT is a medical imaging technique for acquiring high resolution images of the retina and optic nerve. This instrument emits a broad bandwidth, near infrared light from a super-luminescent diode onto the retina. Reflected light rays from the retina are analyzed by interferometry and Fourier-transformed into high resolution quasi-histologic images of the retina and optic nerve.
   4. Slit-Lamp Biomicroscopy Slit-lamp examination of the eyes of all participants will be performed. The slit-lamp utilizes a beam of light and a pair of microscopes to aid in the detailed examination of the ocular tissues from the external parts of the eye, the adnexa, to the posterior aspect including the optic nerve and retina.
   5. Goldman Applanation Tonometry (GAT) Goldman Applanation Tonometry (GAT). Goldman applanation tonometry is a routine test for measuring intraocular pressure (IOP). It is a contact tonometer, therefore, 1 drop of the anesthetic, proparacaine will be used to numb the eye. Two GAT measurements will be taken. If the readings differ by more than 2 mmHg, a third measurement will be carried out. The principal investigator will be masked to the readings. A second optometrist (study optometrist 1) will record the IOPs and the average of two readings with a difference ≤ 2 mmHg will be taken.
   6. Dynamic contour tonometry (DCT) The DCT is a contact tonometer with a concave tip which has an electronic sensor. The radius of curvature of the tip is 10.5 mm. An electronic pressure sensor is integrated into the center of the contacting tip surface. When the tip of the DCT contacts the corneal surface, it conforms to the curvature of the tip. This allows the electronic sensor measure IOP independent of corneal properties. The measured IOP is displayed on the instrument. Two readings with the best quality scores will be averaged and recorded by a study optometrist 1. The principal investigator will be masked to the IOP readings. Intraocular pressure (IOP) measured by most tonometers typically have errors associated with corneal parameters like CCT, CH, and corneal curvature. The DCT will help overcome the influences of these corneal parameters on IOP measurement.
   7. Gonioscopy Gonioscopy is a procedure used to examine the anterior chamber angles of the eye. The procedure is carried out by means of a contact lens called the Gonio lens. Gonioscopy will be performed immediately after GAT. A drop of Proparacaine 1% may be added as needed to prolong local anesthetic effects. Gonioscopy will be used to rule out other forms of glaucoma like Angle closure glaucoma, Inflammatory glaucoma, pigmentary, and pseudo-exfoliation glaucoma.
   8. Dilated Fundus Examination (DFE) Pupillary dilation will be done with the instillation of 1% tropicamide in both eyes. Detailed examination of the anterior chamber, lens, vitreous, optic nerve, macular, retinal up to the periphery of the retina, will be performed. The purpose of the DFE is to establish the baseline ocular status and to rule out ocular diseases that may confound the findings of the study.
   9. Systemic blood pressure (BP) The BP of all participants will be measured using an automatic blood pressure measuring device. The ocular perfusion pressure (OPP) will be calculated by taking the difference of the systolic blood pressure (SBP) and the IOP (OPP = SBP - IOP). Arterial pulse amplitude (APA) will be calculated by taking the difference of the SBP and diastolic BP (DBP) (APA = SBP - DBP).
3. Adherence to treatment

   In order to monitor adherence to treatment, participants will be given a calendar log to write in the number of drops instilled, the date and time of instillation.
4. Follow-up visit schedule:

   Follow-up visits after the onset of treatment will be 2 weeks, 6 weeks, and 3 months after the onset of treatment. Please see below for what data will be collected for these follow-up visits.
5. Procedures to be carried out at follow-up visits The following procedures will be carried out at all the follow-up visits outlined above.

   * Assessment of participants' logbook to ensure adherence to treatment. Level of adherence will be quantified based on the number of drops, and days missed.
   * A traditional paper survey will be used to assess possible adverse events.
   * Slit lamp examination to elicit any signs of adverse events and signs of disease progression.
   * GAT to measure IOPs.
   * ORA to measure CH, CRF, IOPcc, and IOPg.
   * DCT to measure IOP and OPA.
6. Statistical analysis and sample size calculation

   a. Intent-to-treat analyses (ITT) This protocol shall follow the ITT analyses. All participant data shall be analyzed in the original treatment assignment even if they discontinue study mid-way or change treatment assignments.

   Two sample size calculations were performed. The first was for non-inferiority between netarsudil and bimatoprost. The second was for a sub-group analysis of the effect of corneal thickness and CH on the efficacy of both drugs. Since the sub-group analysis yielded the highest sample size, details were presented here. Subjects were classified into 2 CCT sub-groups (thin corneas: ≤ 540 µm, thick: > 540 µm) based on the classification scheme used by Johnson et al (2008). The change in IOP in those with thin corneas treated with netarsudil will be compared to those with thin corneas treated with Lumigan. The same comparison will be made for those with thick corneas. An effect size of 2.4 mmHg was used based on derivation from a SD of 3.0. Assuming a power = 80%, and an alpha = 0.05, the calculated sample size was 26. Since we have 2 groups (thin and thick corneas) with 2 treatment arms (netarsudil and bimatoprost), the total calculated sample size for the 4 groups was 104. A 10% increase was added to the calculated sample size to account for attrition. The total sample size needed to detect the effects of all the aims of research is therefore 115.
7. Data Storage and Confidentiality.

   1. Data Storage:

      Hard copies of data including OCT, Visual field, Ocular Response Analyzer printouts will be collected and kept in the individual participant record folder. All individual record folders will be stored in secure, locked metal cabinets. All digital data will be stored in a password-protected computer. All data will be made available to the Salus University Institutional Review Board (IRB) upon request. The analysis of the data for presentation will only show participants ID and age.
   2. Data management:

   All data shall be kept in the Essential document folder, and pertinent data from all individual participant forms shall be stored in a safe, password-protected computer. All individual participant data will further be aggregated in a spreadsheet, de-identified, and made ready for analysis.
8. RISK/BENEFIT ASSESSMENT

   1. Potential Risks. The risks involved in the intervention are the same risks patients are normally exposed to in clinical practice with the treatment of NTG.

      Expected risks with the use of netarsudil and bimatoprost include conjunctival hyperemia, redness, stinging or burning sensation, and dry eyes. Changes in iris pigmentation could result from the use of bimatoprost.
   2. Risk Classification. The overall risk classification for the study is minimal and not greater than what is normally experienced in clinical practice. This definition of minimal risk is in accordance with the Health and Human Services/Food and Drugs Administration (HHS/FDA) Regulations which classifies minimal risk as "the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests."
   3. Protection Against Risks. The safety of treatment will be assessed at every visit with a patient interview and a thorough eye examination. The study does not have a Data Safety Monitoring Board (DSMB). However, all adverse events will be promptly reported to the Salus University IRB.
   4. Potential Benefits to the Subject. The study protocol involves the treatment of NTG with standard FDA-approved medical treatment for glaucoma. This is necessary to prevent progression of the disease.
   5. Potential Benefits to Society. This project may provide evidence for a more efficacious treatment of NTG. Secondly, it may provide evidence for the adequate control of IOP in NTG patients with thicker corneas, and or greater CH.
9. Therapeutic Alternatives. Many therapeutic alternatives exist for the study participants. These alternatives include, latanoprost, travoprost, latanoprostene bunod, combigan, timolol, dorzolamide, etc. The therapeutic agents used in this study, and other agents will also be available to any participant who chooses not to continue in the study but wishes to continue with the treatment.
10. Risk/Benefit Relationship. netarsudil and bimatoprost have been shown to be efficacious anti-glaucoma agents. These agents are already being widely used in clinical practice. The risks posed by these agents do not exceed that of alternatives. The benefits include reduction of IOPs, and reduction in the risk of progression of glaucoma. The benefits of this study therefore outweigh the potential risks.
11. Financial Compensation for Participation. Subjects who complete the 3 months of follow-up visit will receive a $20 Target gift card.
12. SUBJECT IDENTIFICATION, RECRUITMENT, AND CONSENT Method of Subject Identification and Recruitment. Potential participants will be recruited from patients attending regular clinic at Roberts Eyecare Associates in Vestal New York. Flyers will be designed and handed to other eyecare practices announcing the clinical trial. All potential participants will undergo a complete eye examination to determine their eligibility for inclusion. All those meeting the inclusion criteria will be informed of the study. Those who agree to participate will be given an informed consent form to read. Only those who agree to participate after reading and demonstrating understanding of the entailments of the study and has duly signed, will be recruited.
13. Competing Protocols. After searching the National Institute of Health (NIH) registered clinical trials, at this time, there seem to be no competing protocol with substantial eligibility criteria as this study.
14. Subject Competency. All subjects are expected to be competent to give informed consent. If a subject who meets the eligibility criteria is not competent to give informed consent, an informed consent shall be sought from the participant's legal healthcare proxy.
15. Process of Informed Consent. Informed consent will be sought from all subjects to be recruited for the study. The inform consent will include a detailed explanation of the purpose of the study in a language that is accessible to a fifth-grade student. It will also include an explanation of the risks and benefits of the study interventions. Participants in the study will also be advised of expected adverse events they may experience. They will be informed of their rights to discontinue participation in the study at any time. A statement reassuring participants that treatment for glaucoma will continue even if they choose to leave the study, will also be included in the informed consent form. Only subjects who have received instructions on the study and have signed the informed consent form will be recruited for the study. The informed consent form will be filled at least two weeks before the commencement of the study.

    The consent form shall contain no statement penalizing subjects for non-participation, or statements absolving the study researchers of legal responsibilities in cases of severe adverse events or misconduct.
16. Subject/Representative Comprehension. All subjects or their legal representatives will be asked if they understand the content of the informed consent. If they confirm understanding they will be encouraged to explain, to the best of their understanding, what the study entails, and the content of the formed consent form. This will include, purpose of the study, procedures, potential risks, potential benefits, alternatives, and any other information pertinent to informed consent.
17. Information Purposely Withheld. No information will be purposely withheld from the subject.
18. Documentation of Consent/Assent. Edgar U Ekure (OD, MS, FAAO) shall be responsible for documenting the obtainment of informed consent from the subject.

ELIGIBILITY:
-Inclusion Criteria:

* New NTG patients naïve to treatment.
* Patient with 360 degrees open angles on gonioscopy.
* Patients with glaucomatous optic neuropathies (GON).
* Patients with three repeatable visual field defects over two visits.
* Subjects must have IOPs ≤ 21 mmHg and no recorded IOPs > 21 mmHg at any time.

Glaucomatous optic neuropathy and visual field criteria:

Category 1 and 2 of the glaucoma diagnostic criteria of the International Society of Geographical and Epidemiological Ophthalmology (ISGEO) will be adopted in this study.

ISGEO Category 1 classification of glaucoma:

Reliable and repeatable visual field defects consistent with a glaucomatous optic neuropathy, and either a vertical cup-disc ratio (VCDR) at the 97.5th percentile of the normal population (about 0.7 VCDR), or VCDR asymmetry between the right and left eyes at the 97.5th percentile of the normal population (i.e., about 0.2).

ISGEO Category 2 classification of glaucoma:

Visual field results are not definitive or are unattainable due to patient inability to perform an adequate quality test, and optic disc has VCDR of at the 99.5th percentile of the normal population (i.e., VCDR of about 0.9) or VCDR asymmetry between the right and left eyes at the 99.5th percentile of the normal population (i.e a CDR asymmetry of about 0.3).

-Exclusion Criteria

* Patients with IOPs greater than 21 mmHg at any previous point in time
* Patients with corneal pathology
* Previous ocular surgery in the past 6 months
* Patients with any other types of glaucoma other than NTG
* Patients who are unwilling or unable to follow-up for a 3-month period
* Patients with systemic conditions where a non-glaucomatous optic neuropathy cannot be ruled out.
* Subjects who are pregnant, breastfeeding, or considering becoming pregnant
* Subjects who could be pregnant will be screened for pregnancy thus: Those who are not pregnant nor considering becoming pregnant and are not on any birth-control at the time of recruitment will be excluded from participation because of the risk of pregnancy unknown to the patient at the time of recruitment.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Post-treatment IOP | 3 months post-treatment
  Change in IOPs (GAT, DCT, and ORA) from baseline.

SECONDARY OUTCOMES:
Post-treatment IOP change by CCT | 3 months post-treatment
  Change in IOPs (GAT, DCT, and ORA) from baseline among subjects with thin and thick corneas.
Post-treatment IOP change by CH | 3 months post-treatment
  Change in IOPs (GAT, DCT, and ORA) from baseline among subjects with the lower and higher 50 percentile of CH.
Post-treatment change in CCT | 3 months post-treatment
  Change in CCT from baseline
Post-treatment change in CH | 3 months post-treatment
  Change in CH from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jingyun Wang, Ph.D, Study Director — Salus University
Locations (1):
- Roberts Eyecare Associates, Vestal, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
1. Raw clean data for statistical analyses
  2. Other data will be shared as needed
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months to 1 year after after completion of study
Access Criteria: Access to IPD shall be obtained through email request from Edgar U Ekure (OD, MS, FAAO). Email: exe0003@salus.edu